CLINICAL TRIAL: NCT07385079
Title: A Randomized, Multicenter, Phase 3 Trial of Anlotinib Plus Immunochemoradiotherapy vs Immunochemoradiotherapy in High-Risk Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Anlotinib Plus Immunotherapy and Chemoradiotherapy for High-Risk Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-257-FLK
Record Dates: First submitted 2025-09-23; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Nasopharyngeal Cancinoma (NPC); Nasopharyngeal Cancer
Keywords: anlotinib hydrochloride; PD-L1 antibody; chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anlotinib hydrochloride Arm (Experimental): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), and benmelstobart (1200mg, d1) every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. Anlotinib hydrochloride (10mg, d1-d14) will be given every 3 weeks for 3 cycles in induction chemotherapy. Subsequently, adjuvant therapy with benmelstobart (1200 mg, d1) will be initiated for a total of 9 cycles.
  Interventions: Drug: Anlotinib Hydrochloride Capsules; Drug: Gemcitabine (GEM); Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy; Drug: Benmelstobart
- PD-L1+Chemoradiation Arm (Active Comparator): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), and benmelstobart (1200mg, d1) every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. Adjuvant therapy with benmelstobart (1200 mg, d1) will be initiated for a total of 9 cycles.
  Interventions: Drug: Gemcitabine (GEM); Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy; Drug: Benmelstobart

INTERVENTIONS:
Drug: Anlotinib Hydrochloride Capsules — Anlotinib hydrochloride (10mg, d1-d14) will be given every 3 weeks for 3 cycles in induction chemotherapy.
  Arms: anlotinib hydrochloride Arm
Drug: Gemcitabine (GEM) — Gemcitabine 1g/m2, d1 & 8 of every cycle, every 3 weeks for 3 cycles before radiation.
Drug: Cisplatin — Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation; Concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiation
Radiation: Intensity-modulated radiotherapy — Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy will be given in 33 fractions.
Drug: Benmelstobart — Benmelstobart 1200mg will be given every 3 weeks for 3 cycles in induction chemotherapy and for 9 cycles in adjuvant chemotherapy, started on day 1 of induction chemotherapy and adjuvant chemotherapy, respectively.

SUMMARY:
This trial aimed to evaluate the efficacy of anlotinib hydrochloride combined with benmelstobart, induction chemotherapy, and concurrent chemoradiotherapy (IC+CCRT), versus a regimen of benmelstobart plus IC+CCRT, in patients with high-risk locoregionally advanced nasopharyngeal carcinoma (LANPC).

DETAILED DESCRIPTION:
This trial will enroll patients with locoregionally advanced nasopharyngeal carcinoma (LANPC) staged as T4N2 or T1-4N3 (AJCC 9th edition). Participants will be randomized 1:1 to either the control or experimental regimen. The control regimen consists of three cycles of induction chemotherapy (gemcitabine, cisplatin, and benmelstobart), followed by concurrent cisplatin-based chemoradiotherapy and 9 cycles of benmelstobart as adjuvant therapy. The experimental group will receive the same regimen plus anlotinib hydrochloride during the induction chemotherapy phase. All patients will receive intensity-modulated radiotherapy (IMRT). In the experimental group, anlotinib hydrochloride will be administered on days 1-14 of each 3-week induction cycle for three cycles.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 and ≤65 years
2. Patients with histologically confirmed non-keratinizing nasopharyngeal carcinoma according to WHO criteria.
3. Tumor staged as T4N2 and T1-4N3 (AJCC 9th)
4. Eastern Cooperative Oncology Group performance score of 0-11.
5. Adequate marrow function: white blood cell count > 4 × 10⁹/L hemoglobin >90g/L and platelet count >100×10⁹/L
6. Adequate hepatic and renal function：

   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×ULN
   * Alkaline phosphatase ≤ 2.5 × ULN
   * clearance rate ≥ 60 ml/min
7. Other laboratory and clinical criteria

   * Normal thyroid function, serum amylase and lipase, pituitary hormone levels, inflammatory markers, cardiac enzyme tests and electrocardiogram (ECG)
   * For patients aged >50 years with a history of smoking, normal pulmonary function test (PFT) results are required
   * For patients with abnormal ECG findings or a prior history of cardiovascular disease (not meeting any exclusion criteria listed in Item 8), additional assessments including myocardial function evaluation and cardiac ultrasound (echocardiography) must be performed, with results within normal limits
8. Patients must be informed of the investigational nature of this study and give written informed consent, and be willing and able to comply with the study schedule, including follow-up visits, treatment procedures, laboratory testing, and other protocol-related requirements.
9. Women of childbearing potential (WOCBP) must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug (e.g., condoms, physician-guided regular use of oral contraceptives).

Exclusion Criteria

1. Positive for hepatitis B surface antigen (HBsAg) with hepatitis B virus DNA >1×103 copies/mL, positive for anti-hepatitis C virus (HCV) antibody , positive for anti-hepatitis C virus (HCV) antibody
2. Positive for anti-HIV antibody or diagnosed with acquired immunodeficiency syndrome (AIDS).
3. Active pulmonary tuberculosis: Patients with a history of active tuberculosis within the past year should be excluded regardless of treatment status. Patients with a history of active pulmonary tuberculosis more than one year prior should also be excluded, unless they received confirmed and regular anti-tuberculosis treatment.
4. Active, known, or suspected autoimmune diseases, including but not limited to uveitis, colitis, hepatitis, hypophysitis, nephritis, vasculitis, systemic lupus erythematosus, hyperthyroidism, hypothyroidism, and asthma requiring bronchodilators. Type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) are allowed.
5. History of interstitial lung disease or pneumonia requiring oral or intravenous corticosteroids within the past year; use of vancomycin within the past month.
6. Ongoing chronic systemic corticosteroid therapy (equivalent to or greater than prednisone >10mg per day) or any other immunosuppressive therapy. Patients received inhale or topical corticosteroid are allowed.
7. Uncontrolled cardiac conditions, such as:

   * Heart failure with New York Heart Association (NYHA) classification ≥ Class II;
   * Unstable angina;
   * History of myocardial infarction within the past year;
   * Supraventricular or ventricular arrhythmias requiring treatment or intervention
8. Pregnant or breastfeeding women (pregnancy testing should be considered for women of childbearing potential with active sexual life)
9. History or presence of other malignancies, except for adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, and papillary thyroid carcinoma.
10. Known hypersensitivity to macromolecule protein products or any component of benmelstobart.
11. Active infections requiring systemic treatment within 1 week prior to enrollment.
12. Administration of live vaccines within 30 days prior to the first dose of anlotinib hydrochloride.
13. History of organ transplantation or hematopoietic stem cell transplantation.
14. Presence of clinically significant bleeding symptoms or a definite hemorrhagic tendency; specifically, cases with a high risk of bleeding from local recurrence, or those within one year post-radiotherapy assessed to have a high risk of necrosis, must be excluded.
15. History of hypertension that remains poorly controlled with medication (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg).
16. Urinalysis showing urine protein ≥ ++, confirmed by 24-hour urine protein quantification ≥1.0 g.
17. Factors significantly affecting the absorption of oral drugs, such as inability to swallow, chronic diarrhea, or intestinal obstruction.
18. Any other condition assessed by the investigator as potentially compromising patient safety or compliance, such as severe illnesses requiring urgent treatment (including psychiatric disorders), significantly abnormal laboratory values, or other psychological, familial, or social risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3 year
  From date of randomization until the date of first documented locoregional recurrence, distant metastasis, or death from any cause, whichever occurred first

SECONDARY OUTCOMES:
Tumor response | the time of completion of induction chemotherapy, radiotherapy, and adjuvant immunotherapy; from the date of enrollment until the date of the last time that tumorimaging and assessment of disease has been done, assessed up to 62 weeks
  Evaluation of tumor response as CR, PR, SD, PD, NA by clinicians
Overall survival (OS) | 3 years
  From date of randomization until the date of death from any cause, whichever came first
Distant metastasis-free survival (DMFS) | 3 years
  From date of randomization until the date of first documented distant metastasis, whichever occurred first.
Locoregional recurrence-free survival (LRRFS) | 3 years
  From date of randomization until the date of first documented locoregional recurrence, whichever occurred first.
Adverse events (AEs) and serious adverse events (SAEs) | 3 years
  Graded according to CTCAE V5.0.
Quality of life (QoL) | week 1, 6, 24, 60, 72
  The change of QoL from randomization to the start of radiotherapy, the end of radiotherapy, 13-16 weeks after radiotherapy, 2 years and 3 years after randomization. The EORTC QoL questionnaire-C30 (EORTC QLQ-C30）version 3.0 will be used. This questionnaire comprises 30 questions, 24 of which are aggregated into nine multi-question scales, that is, five functioning scales (e.g., physical), three symptom scales (e.g., fatigue) and one global health status scale. The remaining six single-question (e.g., dyspnoea) scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual. For the functional scales and the global health status scale, a higher score represents a better level of functioning or quality of life. For the symptom scales, a higher score indicates a greater severity of symptoms.
Failure-free survival (FFS) within different subgroups | 3 years
  analyses for FFS will be performed within the following subgroups: Epstein-Barr virus (EBV) DNA (≤4000copies/ml vs. >4000copies/ml), different PD-L1 expression levels, age, gender, performance status, T category, N category, and stage.

OTHER OUTCOMES:
Correlation between pre-treatment PD-L1 expression level and FFS | 3 years
  Pre-treatment PD-L1 expression level of tumor cell is evaluated centrally by means of immunohistochemical testing.
Evaluate failure-free survival in the subgroup of plasma Epstein-Barr virus DNA level | 3 years
  Subgroup analysis
Evaluate failure-free survival in the subgroup of clinical stage | 3 years
  Subgroup analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No
Complete de-identified patient data set will be submitted onto an online platform.